CLINICAL TRIAL: NCT04939311
Title: Immunomodulation Using VB-201 to Reduce Arterial Inflammation in Treated HIV - VITAL HIV Trial
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding for this trial has not been established.
Sponsor: Priscilla Hsue, MD (Other)
Collaborators: University of California, Los Angeles (Other); University of Utah (Other)
Responsible Party: Sponsor-Investigator, Priscilla Hsue, MD, Chief of Cardiology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VITAL HIV
Record Dates: First submitted 2021-06-03; First posted 2021-06-25 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Inflammation; HIV Infection; Cardiovascular Disease
MeSH Terms: conditions — Inflammation; HIV Infections; Cardiovascular Diseases | interventions — 1-palmityl-2-(4-carboxybutyl)-sn-glycero-3-phosphocholine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VB-201 (Experimental): One dose of VB-201 80 mg (1 tablet) will be administered orally once daily for 52 weeks.
  Interventions: Drug: VB-201
- Placebo (Placebo Comparator): One dose of placebo 80 mg (1 tablet) will be administered orally once daily for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VB-201 — One dose of VB-201 80 mg (1 tablet) will be administered orally once daily for 52 weeks.
  Arms: VB-201
Drug: Placebo — One dose of placebo 80 mg (1 tablet) will be administered orally once daily for 52 weeks.
  Arms: Placebo

SUMMARY:
This study is a double blinded, placebo-controlled, randomized, parallel group study, designed to compare the efficacy and safety of VB-201 80mg taken orally once daily to placebo for anti-inflammation in HIV-infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* On continuous antiretroviral therapy and virologically suppressed HIV infection for ≥12 weeks prior to study entry
* CD4 T-cell count > 350 cells/mm3
* Male or female between the ages ≥ 40 years of age to <≤75
* Documented cardiovascular disease (1. Prior myocardial infarction, 2. History of percutaneous coronary intervention, 3. History of coronary artery bypass graft OR 4. Angiographic evidence of >50% stenosis in at least one coronary artery] OR 1 CVD risk factor (T2DM, current smoking, hypertension, dyslipidemia, hsCRP≥2mg/L, family history)
* TBR of >1.6 of the MDS of the carotid/aorta at baseline. This baseline arterial TBR cutoff excludes the rare individual that lacks appreciable arterial inflammation. It is notable that while 5-10% of uninfected individuals will have lower TBRs, it is rare that an HIV infected individual will fall below this range.
* Female subjects must either be of non-childbearing potential as defined by menopause with amenorrhea for >2 years, bilateral oophorectomy, or agree to use adequate contraception throughout the study and for at least one month following termination and have a negative pregnancy test at screening prior to the first dose of drug.
* Males must use at least one method of contraception throughout the study.

Exclusion Criteria:

* Pregnant/nursing women
* Uncontrolled hypertension or diabetes requiring insulin
* AST/ALT or alkaline phosphatase >2x ULN
* Cancer within the last 5 years with exception of squamous cell carcinoma and basal cell carcinoma
* Nephrotic syndrome or eGFR <60 mL/min/1.73m2
* Cytopenias which include 1) WBC <3.5 x103/uL 2) Platelet <120 x103/uL 3) ANC <1.5 x103/uL, and absolute lymphocytes <0.8 x 103/uL
* Anemia as fined by <10 g/dL
* Evidence of tuberculosis infection at screening within 30 days prior to screening.
* Family history of long QT syndrome, using medication that prolongs QT internal, OR evidence of prolonged QT of >470 msec as evidenced by ECG
* Acute systemic infection within 30 days
* On additional immunosuppressant or immunomodulatory therapies

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Target-to-background ratio (TBR) | 1 year (Baseline and Week 52)
  Change in Target-to-background ratio (TBR) from baseline to follow-up study at 52 weeks as assessed by Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography (FDG PET/CT)

SECONDARY OUTCOMES:
Change in high sensitivity C-reactive protein (hs-CRP) in mg/L | 1 year (Change from baseline to week 24 and baseline to week 52)
  Change in hs-CRP from baseline to week 24 and baseline to week 52 as measured by blood collection
Change in Interleukin-6 (IL-6) in pg/mL | 1 year (Change from baseline to week 24 and baseline to week 52)
  Change in IL-6 from baseline to week 24 and baseline to week 52 as measured by blood collection
Change in soluble cluster of differentiation (sCD163) ng/mL | 1 year (Change from baseline to week 24 and baseline to week 52)
  Change in sCD163 from baseline to week 24 and baseline to week 52 as measured by blood collection
Change in Lipoprotein (a) [Lp(a)] in mg/dL | 1 year (Change from baseline to week 24 and baseline to week 52)
  Change in Lp(a) from baseline to week 24 and baseline to week 52 as measured by blood collection
Change in Lipoprotein-associated Phospholipase A2 (Lp-PLA2) in ng/mL | 1 year (Change from baseline to week 24 and baseline to week 52)
  Change in Lp-PLA2 from baseline to week 24 and baseline to week 52 as measured by blood collection
Change in D-Dimer (ng/mL) | 1 year (Change from baseline to week 24 and baseline to week 52)
  Change in D-Dimer from baseline to week 24 and baseline to week 52 as measured by blood collection
Change in Markers of Immune Activation | 1 year (Change from baseline to week 24 and baseline to week 52)
  Change in Co-expression of HLA-DR/CD38 on T-cells from baseline to week 24 and baseline to week 52 as measured by blood collection
Change in Monocyte Activation | 1 year (Change from baseline to week 24 and baseline to week 52)
  Change in Co-expression of CD14/CD16 on Monocytes from baseline to week 24 and baseline to week 52

OTHER OUTCOMES:
Change in non-calcified plaque progression | 1 year (Baseline and Week 52)
  Change in non-calcified plaque progression from baseline to week 52 as assessed by Coronary Computed Tomography Angiography (Coronary CTA)
Change in high risk plaque | 1 year (Baseline and Week 52)
  Change in high-risk plaque from baseline to week 52 as assessed by Coronary Computed Tomography Angiography (Coronary CTA)
Incidence of new lesions | 1 year (Baseline and Week 52)
  Incidence of new lesions from baseline to week 52 as assessed by Coronary Computed Tomography Angiography (Coronary CTA)

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Hsue, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No